CLINICAL TRIAL: NCT07122973
Title: Pain and Itch Neuromodulation: Effects of Offset Analgesia, Placebo, and Nocebo and Topographical Distribution of Itch and Pain Receptors
Brief Title: Topographical Distribution of Itch and Pain Receptors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20250017 Project 4
Record Dates: First submitted 2025-08-13; First posted 2025-08-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pain; Itch
MeSH Terms: conditions — Pain; Pruritus | interventions — Histamine; Capsaicin; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Itch and pain (Experimental)
  Interventions: Other: Histamine; Other: Cowhage; Other: Capsaicin 8% Patch; Other: Demo patch

INTERVENTIONS:
Other: Histamine — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied
Other: Cowhage — The spicules will be manually inserted. Approximately 30-35 spicules are gently rubbed into a 1 cm diameter skin area on the forearm/face
Other: Capsaicin 8% Patch — Capsaicin patches (dosage form: transdermal patch 8% Qutenza, Astellas) will be applied on 3 squared areas in the face.
Other: Demo patch — Placebo patch (demo patch, containing the same formulation as the active treatment with the exception of capsaicin) will be applied on 3 squared areas in the face.

SUMMARY:
The experiment consists of three experimental sessions conducted on three consecutive days.

In all experimental sessions, the participant will fill in a series of questionnaires about how you perceive itch and pain, and about some traits of your personality, such as depression, anxiety and stress.

In the first session, we will mark six test areas in your face (three on each side on jaw, cheek, and temple, respectively). Thent a series of measure-ments in each test area will be conducted:measurement of the blood flow in the skin and sensitivity tests to pressure, pinprick and stroke with a brush.

In the second session, histamine will be applied in one side of the face. On the other side, cowhage spicules will be applied. After 10 minutes, all the tests will be conducted again.

The third session will be identical to the second. However, instead of histamine and spicules, patches containing capsaicin will be applied. In the other side, we will apply patches with placebo (i.e., a non-active patch). After 20 minutes all the tests will be conducted again.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other drugs
* Previous or current history of neurological, immunological, musculoskeletal, cardiac disorder or psychiatric diagnoses that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia, etc.)
* Moles, wounds, scars, or tattoos in the area to be treated or tested
* Current use of medications that may affect the trial such as antihistamines and pain killers
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain and itch
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical studies)
* Contraindications to capsaicin, including intolerance to chili or burns or wounds at the application site
* The subject is assessed as unable to engage in the necessary cooperation required by the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring pain by computerized Visual Analog Scale Scoring | Baseline
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Measuring itch by computerized Visual Analog Scale Scoring | Baseline
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Measuring pain by computerized Visual Analog Scale Scoring | Immediately after the intervention
  We will ask the subjects to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Measuring itch by computerized Visual Analog Scale Scoring | Immediately after the intervention
  We will ask the subjects to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".

SECONDARY OUTCOMES:
Superficial blood perfusion | Baseline
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Superficial blood perfusion | Immediately after the intervention
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Alloknesis | Baseline
  Measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Alloknesis | Immediately after the intervention
  Measured using a standardized sensory brush exerting a force of 200 to 400 mN.
Mechanically evoked itch (MEI) | Baseline
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanically evoked itch (MEI) | Immediately after the intervention
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanical Pain Thresholds (MPT) | Baseline
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Thresholds (MPT) | Immediately after the intervention
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS) | Baseline
  This test is conducted with the same pinprick set used to test the MPT.
Mechanical Pain Sensitivity (MPS) | Immediately after the intervention
  This test is conducted with the same pinprick set used to test the MPT.
Cold Detection Thresholds (CDT) | Baseline
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Thresholds (CDT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Baseline
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Baseline
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Baseline
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thresholds (HPT) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Baseline
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Immediately after the intervention
  The tests of thermal sensation will all be conducted using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain Catastrophizing Scale (PCS). | Baseline
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Itch Catastrophizing Scale (ICS). | Baseline
  The ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Learned Helplessness Scale (LHS) | Baseline
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Learned Helplessness Scale (LHS) | 10 minutes after every induction
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Pain Catastrophizing Scale (PCS). | 10 minutes after induction
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Itch Catastrophizing Scale (ICS). | 10 minutes after induction
  The ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Depression, Anxiety, Stress Scale (DASS-21) | Baseline
  The questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much"
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | Baseline
  The RST-PQ contains in total, 65 items must be answered on a 4-point Likert-type scale
Difficulties in Emotion Regulation Scale Short Form (DERS-SF) | Baseline
  The questionnaire is an 18-item measure used to identify emotional regulation issues in adults. Participants rate each item on a 5-point Likert scale (from 1 to 5).
Emotion Regulation Questionnaire (ERQ | Baseline
  This questionnaire is designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree), where 4 means (neutral).

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Aalborg, Denmark